CLINICAL TRIAL: NCT03091803
Title: Evaluation of Regional Gadolinium Retention in the Brain Using QSM With Correlation to Regional DCE MRI Permeability Using GOCART Technique in Intracranial Neoplasm Patients Receiving Gadobenate Dimeglumine (MultiHance) or Gadoterate Meglumine (Dotarem)
Brief Title: QSM and Regional DCE MRI Permeability Using GOCART Technique
Status: Withdrawn | Type: Observational
Why Stopped: No accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6B-16-1; NCI-2017-00499 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6B-16-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging; gadobenic acid; gadoterate meglumine; gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Arm I (QSM, T1WI, gadobenate dimeglumine, GOCART DCE MRI): Patients undergo standard of care QSM and T1WI. Patients then receive gadobenate dimeglumine IV and undergo GOCART DCE MRI over 60 minutes.
  Interventions: Device: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Gadobenate Dimeglumine; Device: Magnetic Resonance Imaging
- Arm II (QSM, T1WI, gadoterate meglumine, GOCART DCE MRI): Patients undergo standard of care QSM and T1WI. Patients then receive gadoterate meglumine IV and undergo GOCART DCE MRI over 60 minutes.
  Interventions: Device: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Gadoterate Meglumine; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo GOCART DCE MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Drug: Gadobenate Dimeglumine — Given IV
  Other Names: Gd-BOPTA; MultiHance
  Groups: Arm I (QSM, T1WI, gadobenate dimeglumine, GOCART DCE MRI)
Drug: Gadoterate Meglumine — Given IV
  Other Names: DOTAREM; Gd-DOTA
  Groups: Arm II (QSM, T1WI, gadoterate meglumine, GOCART DCE MRI)
Device: Magnetic Resonance Imaging — Undergo QSM and T1WI imaging
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This randomized pilot clinical trial studies quantitative susceptibility mapping (QSM) and regional dynamic contrast enhanced (DCE) magnetic resonance imaging (MRI) permeability using golden-angle cartesian randomized time-resolved (GOCART) technique in evaluating regional gadolinium retention in the brain in patients with intracranial neoplasm receiving gadobenate dimeglumine or gadoterate meglumine. MRI diagnostic techniques such as, QSM and DCE MRI, may help to gather information regarding brain changes associated with gadolinium deposits during 8 to 18 months after administration of gadobenate dimeglumine or gadoterate meglumine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data (e.g. mean, variance, distribution) in the regional brain parenchymal changes associated with gadolinium (Gd) deposition during 8 to 18 months period after administration of gadolinium based contrast agents (GBCA) to Gd naive intracranial neoplasm patients who will be randomized to gadobenate dimeglumine (MultiHance) or gadoterate meglumine (Dotarem).

II. To explore if areas of increased regional Gd deposition at individual level are correlated with baseline regional DCE permeability metrics such as volume transfer coefficient reflecting vascular permeability (kTrans), extracellular volume ratio reflecting vascular permeability (ve) and plasma volume (vp) in intracranial neoplasm patients.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard of care QSM and T1 weighted imaging (T1WI). Patients then receive gadobenate dimeglumine intravenously (IV) and undergo GOCART DCE MRI over 60 minutes.

ARM II: Patients undergo standard of care QSM and T1WI. Patients then receive gadoterate meglumine IV and undergo GOCART DCE MRI over 60 minutes.

After completion of study, patients are followed up at 8-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected intracranial neoplasm scheduled for routine MRI with GBCA (gadolinium naive patients)
* Willingness to comply with the study protocol

Exclusion Criteria:

* Contraindications for MRI or GBCA (standard of care)
* Abnormal renal function with estimated glomerular filtration rate (eGFR) less than 30 mL/min/m^2 based on creatinine obtained within last 30 days
* History of previous administration of GBCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at USC/Norris Comprehensive Cancer Center who are found to have suspected intracranial neoplasm scheduled for routine MRI with GBCA (gadolinium naive patients) will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-04-04 (Estimated); Study Completion 2021-04-04 (Estimated)

PRIMARY OUTCOMES:
Change in QSM score | Baseline up to 18 months
  Descriptive statistics will be used to describe the magnitude of Gd deposition measured by QSM score in each of the two study groups. Histograms will be generated for QSM score at each time point as well as the change from the baseline for each group. The descriptive statistics will be used to calculate the mean, median, interquartile range, and standard deviation. Box plot and overlying histogram will be used to illustrate the distribution of change in Gd deposition between gadobenate dimeglumine and gadoterate meglumine group. Correlation between QSM score versus (vs.) kTrans and QSM score v

SECONDARY OUTCOMES:
Change in T1WI signal intensity ratio | Baseline up to 18 months
  Descriptive statistics will be used to describe the magnitude of Gd deposition measured by T1WI signal intensity ratio in each of the two study groups. Histograms will be generated for T1WI signal intensity ratio score at each time point as well as the change from the baseline for each group. The descriptive statistics will be used to calculate the mean, median, interquartile range, and standard deviation. Box plot and overlying histogram will be used to illustrate the distribution of change in Gd deposition between gadobenate dimeglumine and gadoterate meglumine group. Correlation between T1W
kTrans and Ve signal using GOCART 3D MRI | Up to 18 months
  The signal (kTrans and Ve) will be obtained in voxel level then taking average within the region of interest (ROI). ROI will be placed on the pons, bilateral globi pallidi, thalami and dentate nuclei to obtain the average signal within the ROI. Averages of all bilateral measurements will be used to calculate the final signal for kTrans and Ve. The final kTrans and Ve signal will only be used to assess the correlation with QSM and T1WI signal intensity ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lerner, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States